CLINICAL TRIAL: NCT05720247
Title: Brief Intervention and Fibroscan for Harmful Drinkers Presenting to the Emergency Department.
Acronym: IBAFiRST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19AE001
Record Dates: First submitted 2022-09-30; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Emergency Department; Fibroscan; Brief Intervention; Screening, Brief Intervention, referral to Treatment (SBIRT)
MeSH Terms: conditions — Alcoholism; Emergencies | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Research collecting outcome data is blinded to the study allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibroscan (Experimental): Screening and brief intervention with additional Fibroscan procedure and sharing of results with patient
  Interventions: Diagnostic Test: Fibroscan; Behavioral: Brief Intervention
- Standard Care (Active Comparator): Screening and brief intervention without Fibroscan
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Diagnostic Test: Fibroscan — Fibroscan is a safe and effective test using ultrasound to measure liver elasticity and can detect early signs of liver disease even before a patient shows symptoms.
  Arms: Fibroscan
Behavioral: Brief Intervention — Short counselling session to discuss drinking behavior, risks to health and available sources of treatment and support.

SUMMARY:
The investigators plan to assess the feasibility of a randomised controlled trial of an innovative screening (Identification), Brief Intervention, Fibroscan and Self-Referral for Specialist Treatment (IBAFiRST) programme for high risk drinkers in the Emergency Department (ED). IBAFiRST extends existing screening and advice given to people with potential alcohol use disorders (AUD) in ED. Currently patients who drink heavily have brief advice and are asked to refer themselves to community specialist alcohol treatment services (ATS) after leaving ED. A Fibroscan is a safe, quick and reliable ultrasound test to see if there are signs of "stiffening" of the liver which can indicate early liver damage. It is recommended as a non-invasive test by the National Institute for Health and Care Excellence (NICE) but is not known to be used within EDs in the UK. The investigators wish to test whether giving the patients the results of this scan will make them more likely to self-refer to ATS. Currently take up rates of ATS are low in this population and too few people are seeking treatment to help them reduce their alcohol intake. Because so little is known about self-referral in ED the investigators are completing a feasibility study before seeking funding for a large scale randomised trial.

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) poses a significant burden to individuals, the population and the health and social care system in the United Kingdom (UK). Chronic liver disease is now the third most common cause of death and costs the National Health Service (NHS) an estimated £3.5 billion per year. This equates to 3.6% of the total NHS budget. The only effective way to reduce the risk of liver damage for people at high risk is to abstain from drinking alcohol. Alcohol services can successfully help people reduce their risk of liver damage by helping them reduce or stop drinking. Many people with AUD use emergency departments and it is NHS policy for them to be screened for harmful drinking and referred for treatment if indicated.

There is currently very little evidence that existing methods to screen for alcohol use disorders and encourage high risk patients to refer themselves to ATS from ED, are effective. Fibroscan is a safe and effective test to look for early signs of liver disease even before a patient shows symptoms. Research into the use of Fibroscan as part of a brief advice intervention for AUDs in ED has not been undertaken before. If effective in increasing treatment uptake the reduction in liver disease from treating more ED attenders could be substantial.

All patients attending the Emergency Department are already asked a single alcohol screening question as part of their normal assessment: "Have you drunk more than 6 units of alcohol on one occasion in the previous month?". Those answering yes are briefly counselled about their alcohol use ( standard brief intervention) and advised to self-refer for community treatment services. During the study these patients will be offered participation in the trial. If they consent the research team will assess their eligibility by using the AUDIT-C questionnaire a widely used set of 6 questions taking approximately 5 minutes to complete. Patients scoring 10 or less will receive a brief intervention and advice on self-referral as usual. Patients scoring 11 or 12 will be eligible to be randomised to a Fibroscan (intervention arm) in addition to brief advice and information (control arm).

All patients will receive the same verbal and printed information about community alcohol treatment services and how to self-refer. Patients will be followed up at 1, 3 and 6 months post randomisation by telephone. A research nurse blinded to the allocation will collect data on their drinking behaviour in the previous week and ask whether they have sought help from alcohol services their General Practitioner (GP) or from other NHS services. In addition the primary outcome measure, engagement in alcohol treatment services at 6 months, will be confirmed by collecting data from the services themselves under a research information sharing agreement. This activity is explained clearly in the information and consent processes for patients given the sensitivity of the information. Study data will be analysed using descriptive statistics and cross-tabulations. This will provide the detailed information necessary to assess the success of the feasibility trial and to inform a power calculation for a full-scale randomised trial of the effect of the Fibroscan intervention in ED.

ELIGIBILITY:
Inclusion Criteria:

* Has capacity to give informed consent
* Have no urgent or life-threatening illness or injury
* Have not eaten a larger meal within 3 hours of trial enrollment
* Answer "yes" to a single item alcohol screening question (standard care)
* Score of 11 or 12 on the Audit-C alcohol screening tool

Exclusion Criteria:

* They are unable or unwilling to undertake single-question screening (standard care)
* They refuse or lack capacity to give informed consent to trial inclusion
* They are living in postcodes outside of the catchment areas for Nottingham City or Nottingham County community alcohol treatment services
* They have an urgent or life-threatening illness or injury
* Their treating clinician thinks there is any other reason that they would not benefit from trial inclusion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As expressed by the patient
Enrollment: 80 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2023-09-23 (Estimated)

PRIMARY OUTCOMES:
Self-referral to community alcohol treatment services | 6 months
  independently confirmed record of self-referral

SECONDARY OUTCOMES:
Alcohol use disorders identification test consumption (AUDIT C) | Baseline, 1, 3 and 6 months
  standardised alcohol risk score
Drinks consumed in previous 7 days | Baseline, 1, 3 and 6 months
  Number of drinks consumed
Days drinking alcohol in the previous 7 days | Baseline, 1, 3 and 6 months
  Days on which any alcohol was consumed
Attendance at an Emergency Department | Baseline, 1, 3 and 6 months
  ED attendance since previous study event

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom